CLINICAL TRIAL: NCT00821184
Title: A Prospective Randomized Trial of Behavioral Modification and Solifenacin (Vesicare)vs Solifenacin (Vesicare) Alone for the Treatment of Urge Incontinence in Patients With an Overactive Bladder
Brief Title: Behavioral Modification and Vesicare Versus Vesicare Alone for Urge Incontinence in Patients With Overactive Bladder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient subject availability/findings for data analysis
Sponsor: Lahey Clinic (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Linda Topjian, Study Coordinator, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-083
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Overactive Bladder
Keywords: urinary incontinence; overactive bladder; urinary frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vesicare (Active Comparator): Vesicare alone
  Interventions: Drug: Vesicare (solifenacin)
- Vesicare/behavioral modification (Active Comparator): Vesicare plus behavioral modification
  Interventions: Behavioral: Vesicare (solifenacin) plus behavioral modification

INTERVENTIONS:
Drug: Vesicare (solifenacin) — 5mg po qd
  Arms: Vesicare
Behavioral: Vesicare (solifenacin) plus behavioral modification — 5 mg dose po once daily plus behavioral modification
  Other Names: Vesicare (solifenacin)
  Arms: Vesicare/behavioral modification

SUMMARY:
This study will help determine if behavior modification performed in conjunction with oral Vesicare anticholinergic therapy is more effective for treating overactive bladder symptoms than oral Vesicare anticholinergic therapy alone.

DETAILED DESCRIPTION:
Overactive bladder symptoms are commonly treated with oral anticholinergic medications that work by stopping muscles from tightening or behavioral modification. This study will help determine if behavior modification (fluid regulation, pelvic exercises, timed voiding) performed in conjunction wth oral Vesicare anticholinergic therapy, is more effective for treating overactive bladder symptoms than oral Vesicare anticholinergic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years of age
* OAB symptoms for > 3 months
* Symptoms defined as greater than 3 episodes/week of an uncontrolled urge to void causing incontinence.
* May or may not be accompanied by urinary frequency
* May be accompanied by stress urinary incontinence where stress incontinence does not predominate

Exclusion Criteria:

* Male Patients
* Underlying cortical or spinal cord pathology including SCI, MS, or
* Parkinson's Disease
* Urinary retention with post-void residual > 150cc
* Current treatment or treatment within the last 3 months with anticholinergic medications
* Patients not able to complete the questionaires or voiding diaries in English
* Pregnancy
* Active urinary tract infections
* Bladder Cancer or unevaluated hematuria
* Known diagnosis of narrow angle glaucoma
* Severe constipation
* History of reduced renal function (CrCl<30ml/min)
* History of liver disease
* Current treatment with cytochrome P450 inhibitor medications

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T Stoffel, M.D., Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vesicare Alone: Vesicare alone in treatment of incontinence
- Vesicare Plus Behavioral Modification: Vesicare plus behavioral modification for treatment of incontinence
Period: Overall Study
Arm/Group | Vesicare Alone | Vesicare Plus Behavioral Modification
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vesicare Alone | Vesicare Plus Behavioral Modification | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Incontinence Episodes Per 24 Hours Measured by Voiding Diaries.
Time Frame: 0 week - 12 weeks
Measure: Mean (Full Range); unit: incontinence episodes per 24 hours
Arm/Group | Vesicare Alone | Vesicare Plus Behavioral Modification
Number analyzed (Participants) | 6 | 6
incontinence episodes per 24 hours | 1 [0 to 5] | 10 [2 to 22]

2. Secondary Outcome: Improvement of Symptom Severity
Time Frame: 3 months
Population: data were not collected
Arm/Group | Vesicare | Vesicare/Behavioral Modification
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vesicare Alone | Vesicare Plus Behavioral Modification
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No